CLINICAL TRIAL: NCT01377675
Title: Assessment of an Interactive Education Tool to Disseminate Best Practice Recommendations on Chronic Obstructive Pulmonary Disease to Primary Care
Brief Title: Web-based, Interactive Professional Education for Chronic Obstructive Pulmonary Disease
Acronym: WipeCOPD
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: American College of Chest Physicians (Other)
Responsible Party: Sponsor
Other Study IDs: WipeCOPD
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Education of Primary Care Clinicians
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Usual curriculum education program: Third year internal medicine residents
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — The third year internal medicine residents completed the usual curriculum for COPD and took one pretest and two posttests to validate the questions.

SUMMARY:
This study involves the development and evaluation of a web-based, interactive education program on chronic obstructive pulmonary disease (COPD) for primary care clinicians.

The research questions that this proposal addresses include:

1. Can an interactive, web-based COPD course be developed to disseminate evidence-based, best practice recommendations to primary care clinicians?
2. Can assessment tools be developed to evaluate the impact of the program on clinician behavior in clinical practice and on patient care?

ELIGIBILITY:
Inclusion Criteria:

* Primary care clinicians in training
* willing to participate

Exclusion Criteria:

* Specialists

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Third year internal medicine residents
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in clinical practice | 9 months

SECONDARY OUTCOMES:
Clinician knowledge and comprehension | 9 months
Clinician self-confidence | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States